CLINICAL TRIAL: NCT04934319
Title: Association Between Balance and the Integrity of Cerebellar White Matter Tracts in a Healthy Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Youngkook Kim, Assistant Professor, The Catholic University of Korea
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: SC20FISI0152
Record Dates: First submitted 2021-06-07; First posted 2021-06-22 (Actual); Last update posted 2022-06-13 (Actual); Status verified 2022-06

CONDITIONS: Balance; Cerebellum
Keywords: Balance; Cerebellum; White matter tract; Diffusion Tensor Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Balance training (Experimental): A single training group
  Interventions: Behavioral: Balance and Proprioceptive Training

INTERVENTIONS:
Behavioral: Balance and Proprioceptive Training — * Step-by-step training (5 levels)
  * 30 minute per training
  * 3 times per week
  * Four weeks

SUMMARY:
The cerebellum is involved in regulating balance and walking and plays a crucial role in the locomotor adaptation and learning processes. This study aims to investigate the association between balance and the integrity of the cerebellar white matter tracts in a healthy population. Healthy participants will undergo four weeks of balance training. The investigators will analyze changes in the microstructural integrity of the cerebellar white matter tract before and after four weeks of balance training.

DETAILED DESCRIPTION:
The cerebellum is involved in regulating balance and walking and plays a crucial role in the locomotor adaptation and learning processes. The cerebellum's intermediate zone, which receives afferent stimuli from the sensorimotor cortex (via the cortico-ponto-cerebellar tract) and peripheral muscles (via the dorsal spinocerebellar tract), contributes to maintaining body posture and regulating walking. Proprioceptive information from the peripheral muscles passes through the dorsal spinocerebellar tract, enters the ipsilateral cerebellar hemisphere via the inferior cerebellar peduncle, and finally projects to the contralateral motor cortex through the cerebello-thalamo-cortical pathways.

Diffusion tensor imaging (DTI) enables microstructural evaluation of the white matter tracts. Both diffusion tensor tractography, to determine the structural connectivity of the whole tract, and DTI-derived parameters, to determine the microstructural organization, can represent the integrity of the cerebellar white matter tracts.

The investigators will evaluate the motor-related white matter tracts, including the corticospinal tract, the cortico-ponto-cerebellar tract, the dorsal spinocerebellar tract, and the dentato-rubro-thalamo-cortical tract. Healthy participants will perform the four weeks of balance training, and DTI will be acquired before and after exercise. The investigators will analyze the DTI-derived parameters of the relevant white matter tracts and analyze the longitudinal changes. The investigators hypothesized that the four weeks of balance training would enhance the integrity of the cerebellar white matter tracts.

ELIGIBILITY:
Inclusion Criteria:

* Mini-mental state examination >=26
* Independent outdoor ambulator

Exclusion Criteria:

* Men/women with any metal implants in their body
* A prior history of psychopathology or a neurological disorders
* A prior history of osteoporosis, advanced osteoarthritis (K-L grade >=3), surgical history of hip or knee arthroplasty
* If any structural abnormalities are detected on their scan

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2021-05-24 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Fractional anisotropy of the cerebellar white matter tracts | Four weeks
  Measurement of the change of DTI-derived parameters before and after balance and proprioceptive training
  1. Tracts of interest
     * Corticospinal tract (CST)
     * Cortico-ponto-cerebellar tract (CPCT)
     * Dentato-rubro-thalamo-cortical tract (DRTCT)
     * Dorsal spinocerebellar tract (DSCT)
  2. Measurement of DTI-derived parameter
     * Fractional anisotropy (FA) values of the CST, CPCT, DRTCT, and DSCT
  3. Units and scoring of the Measurement
     * FA
       * No unit.
       * The measurement ranges from 0 to 1
       * Higher scores indicate better microstructural integrity.
Community Balance & Mobility Scale | Four weeks
  Performance measure before and after balance and proprioceptive training
  1. Measurement
     * 13 domain
     * Unilateral stance, Tandem walking, 180° tandem pivot, Lateral foot scooting, Hopping forward, Crouch and walk, Lateral dodging, Walking & looking, Running with controlled stop, Forward to backward walking, Walk look and carry, Descending stairs, Step-ups x 1 step
  2. Scoring of the Measurement
     * No units.
     * The measurement ranges from 0 to 96
     * Higher scores indicate better postural balance and mobility.

SECONDARY OUTCOMES:
Mean diffusivity of the cerebellar white matter tracts | Four weeks
  Measurement of the change of DTI-derived parameters before and after balance and proprioceptive training
  1. Tracts of interest
     * CST
     * CPCT
     * DRTCT
     * DSCT
  2. Measurement of DTI-derived parameter
     * Mean Diffusivity (MD) values of the CST, CPCT, DRTCT, and DSCT
  3. Units and scoring of the Measurement
     * MD
       * mm^2/second
       * There is no limit on the range (usually ranges 0.00005 - 0.0001 mm^2/second).
       * Higher scores indicate worse microstructural integrity.
Tract volume of the cerebellar white matter tracts | Four weeks
  Measurement of the change of DTI-derived parameters before and after balance and proprioceptive training
  1. Tracts of interest
     * CST
     * CPCT
     * DRTCT
     * DSCT
  2. Measurement of DTI-derived parameter
     * Tract volume (TV) values of the CST, CPCT, DRTCT, and DSCT
  3. Units and scoring of the Measurement
     * TV
       * mm^3
       * There is no limit on the range.
       * Higher scores indicate better microstructural integrity.

CONTACTS AND LOCATIONS:
Overall Officials: Youngkook Kim, Ph.D., Principal Investigator — Yeouido St. Mary's Hospital, College of Medicine, The Catholic University of Korea
Locations (1):
- Yeouido St. Mary's Hospital, Seoul, Yeongdeungpo-gu, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim JS, Kim SH, Lim SH, Im S, Hong BY, Oh J, Kim Y. Degeneration of the Inferior Cerebellar Peduncle After Middle Cerebral Artery Stroke: Another Perspective on Crossed Cerebellar Diaschisis. Stroke. 2019 Oct;50(10):2700-2707. doi: 10.1161/STROKEAHA.119.025723. Epub 2019 Aug 26. PMID 31446886
- [Background] Kim Y, Kim SH, Kim JS, Hong BY. Modification of Cerebellar Afferent Pathway in the Subacute Phase of Stroke. J Stroke Cerebrovasc Dis. 2018 Sep;27(9):2445-2452. doi: 10.1016/j.jstrokecerebrovasdis.2018.04.039. Epub 2018 May 22. PMID 29801815
- [Background] Kim Y, Im S, Kim SH, Park GY. Laterality of cerebellar afferent and efferent pathways in a healthy right-handed population: A diffusion tensor imaging study. J Neurosci Res. 2019 May;97(5):582-596. doi: 10.1002/jnr.24378. Epub 2018 Dec 24. PMID 30582195